CLINICAL TRIAL: NCT00222950
Title: Concentrations of Plant Sterols in Serum and Aortic Valve Cusps: a Prospectiv Observational Study
Brief Title: Concentration of Plant Sterols in Serum and Aortic Valve Cusps
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Other Study IDs: Plant Sterols 159/04; 159/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Aortic Valve Stenosis
Keywords: plant sterols, serum, aortic valve cusps
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study investigates the effect of margarines supplemented with plant sterol esters on serum and cardiovascular tissue concentrations of plant sterols. We assume that consumption of margarine supplemented with plant sterol esters increases serum and cardiovascular tissue concentrations of plant sterols (sitosterol; campesterol).

DETAILED DESCRIPTION:
The role of plant sterols in cardiovascular diseases is controversially debated. There is an increasing body of evidence that indicates that increased plant sterol serum concentrations are correlated with an increased cardiovascular risk. Functional foods such as margarines supplemented with plant sterol esters are advertised to patients with hypercholesterolemia. Numerous studies show that margarines supplemented with plant sterol esters reduce serum cholesterol concentrations significantly. However, there are no studies available investigating relevant clinical endpoints. Nor are there any studies availabe investigating the effect of the consumption of margarines supplemented with plant sterol esters on serum and cardiovascular tissue concentrations. This study is done to investigate the effect of margarines supplemented with plant sterol esters on serum and cardiovascular tissue concentrations.

ELIGIBILITY:
Inclusion Criteria: aortic valve stenosis -

Exclusion Criteria:familial hypercholesterolemia.

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bohm, Professor, Principal Investigator — University of the Saarland
Locations (1):
- University of the Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Derived] Weingartner O, Lutjohann D, Ji S, Weisshoff N, List F, Sudhop T, von Bergmann K, Gertz K, Konig J, Schafers HJ, Endres M, Bohm M, Laufs U. Vascular effects of diet supplementation with plant sterols. J Am Coll Cardiol. 2008 Apr 22;51(16):1553-61. doi: 10.1016/j.jacc.2007.09.074. PMID 18420097